CLINICAL TRIAL: NCT06171919
Title: Improving HIV Care Continuum Outcomes Among Formerly Incarcerated Individuals Through Critical Time Legal Interventions
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Central Florida (Other)
Collaborators: University of Miami (Other); National Institute of Mental Health (NIMH) (NIH); Hope and Help Center of Central Florida Incorporated (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00006010; 3P30MH133399-01S2 (NIH)
Record Dates: First submitted 2023-11-04; First posted 2023-12-15 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: HIV
Keywords: HIV; Care; Incarcerated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CTI-MLP approach (Experimental): To finalize protocols and a medical-legal partnership training manual for health and social service providers at Hope and Help Inc.
  Interventions: Other: Organizational Partnerships
- CTI-MLP assessment (Experimental): To assess the feasibility and acceptability of a comprehensive critical-time intervention medical legal partnership (CTI-MLP) approach to improve HIV care continuum outcomes among formerly incarcerated individuals and determine the most efficient mechanisms for CTI-MLP delivery
  Interventions: Other: HIV Continuum Care

INTERVENTIONS:
Other: Organizational Partnerships — Component 1 is a comprehensive training for all MLP care providers delivered to clinical, social and behavioral, and legal staff to establish a collaborative environment. Component 2 consists of the screening tool and screening protocol that is designed to identify health-harming legal needs and risks of formerly incarcerated individuals living with HIV. Component 3 includes the provision of legal support.
  Arms: CTI-MLP approach
Other: HIV Continuum Care — Participants will be included in the pilot trial. The investigative team will work with the staff at Hope and Help Inc. to identify and recruit those out of care through reviewing electronic medical records.
  Arms: CTI-MLP assessment

SUMMARY:
The purpose of this research is to better understand the impact of receiving legal aid on HIV care continuum outcomes among formerly incarcerated individuals. In addition, the investigators would like to assess the effectiveness of a comprehensive training for providers in increasing knowledge about medical legal partnerships and improving clinic level outcomes, including communication among providers. The training includes several topics including health disparities impacting formerly incarcerated individuals, health-harming legal needs and risks, screening for health-harming legal needs and risks, medical-legal partnership structure and operations, prerequisites for MLPs, embedding legal expertise within regularized case management, co-location of legal services, and data collection and analysis.

DETAILED DESCRIPTION:
Formerly incarcerated individuals are impacted by health-harming legal needs and risks, including lack of access to HIV care, unsafe housing safety, unstable employment, and other issues that often disrupt HIV care. Providing access to legal services can address barriers to HIV care and improve HIV care continuum outcomes for formerly incarcerated individuals. The proposed study, led by the University of Central Florida (Hispanic Serving Institution), together with the University of Miami, and Hope and Help Inc., aims to pilot test a comprehensive critical-time intervention medical legal partnership (CTI-MLP) approach to optimize timely HIV linkage, retention and viral suppression among formerly incarcerated individuals. MLPs have been used by social justice-oriented medical, health, social, and legal service practices to identify and address health-harming legal needs and risks that create barriers to treatment, care, and recovery for several health conditions. MLPs offer an integrated structural intervention that could improve HIV care continuum and psychosocial outcomes among formerly incarcerated individuals. Our CTI-MLP intervention package consists of: 1) training for all MLP staff (clinical, social and behavioral services, and legal) on HIV continuum of care, health-harming legal needs and risks impacting formerly incarcerated individuals, and MLP structure and operations to ensure that an integrated and collaborative environment is established from the earliest stages of the program; 2) training for case managers and court advocate on the legal continuum of care; 3) embedding of legal expertise within regularized case management team meetings; 4) co-locating legal services in health care agencies through MLP inter-organizational partnership; and 5) tailoring and implementing organizational best-practices in communication and information-sharing protocols among providers within MLP, anchored in patient autonomy and choice. In year 1, the investigators will engage a local community advisory board, scientific advisory board, and legal expert panel to finalize protocols and the Medical Legal Partnership Training Manual. In year 2, the investigators will implement the training and pilot test a CTI-MLP initiative with formerly incarcerated individuals living with HIV (n=100). Over a 6-month period, the team will collect (1) patients' health and functioning, including overall physical health, mental health, social health, pain, fatigue, and overall perceived quality of life; (2) data on legal needs and risk factors; (3) patient HIV care clinical outcomes; and (4) clinic-level indicators, including provider-patient communication and readiness for continued implementation and sustainability. The study will be guided by Reach, Effectiveness, Adoption, Implementation, and Maintenance and Consolidated Framework for Implementation Research frameworks. Active engagement will ensure the effective translation and dissemination of our findings into practice. Completion this project will result in an innovative, evidence-based, community driven structural intervention to improve HIV care continuum outcomes among formerly incarcerated individuals.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Living with HIV (as confirmed by medical record)
* HIV viral load of more than 200 copies/mL (as confirmed by medical record)
* Report history of incarceration
* Willing and able to consent to participate in the trial (including accessing their medical records at the health care organization)
* No intent to relocate within the 6 months following their enrollment in the study.

Exclusion Criteria:

* Individuals who self-report having been sentenced to serve under state or federal custody, with a sentence to begin within 6 months from proposed enrollment in the study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-10-12 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
HIV viral load using polymerase chain reaction (PCR) | 1 year
  HIV viral load through HIV Nucleic Acid Amplification Test (NAAT) HIV by PCR HIV RNA Test
HIV linkage and retention and antiretroviral therapy adherence using surveys | 1 year

SECONDARY OUTCOMES:
Quality of Life checklist | 1 year
  A 36-item health questionnaire. It has 8 scales which provide a profile of functionally participant and welfare. The scales contain two general measures, the PCS (Physical Health Component Summary), and MCS (Mental Health Component Summary).
Mental health indicators survey | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- University of Central Florida, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No